CLINICAL TRIAL: NCT06342570
Title: Quantitative Analysis of EEG Changes in Response to Nociception
Status: Recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0462
Record Dates: First submitted 2024-03-13; First posted 2024-04-02 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Patients Undergoing Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- There is no group to describe.: There is no group to describe.
  Interventions: Other: There is no Intervention name to describe.

INTERVENTIONS:
Other: There is no Intervention name to describe. — There is no Intervention name to describe.

SUMMARY:
This study will quantify the nociception using Analgesia Nociception Index (ANI) during general anesthesia and analyze the differences in EEG depending on the degree of nociception. Additionally, the investigators will quantify the nociception during recovery and analyze the differences in EEG depending on the degree of nociception.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged ≥ 19 undergoing laparoscopic surgery

Exclusion Criteria:

* Patients with arrhythmia
* Patients with pacemaker implantation
* Patients who have received a heart transplant
* Patients taking medications that may affect ANI (antimuscarinics, alpha-agonist, beta blockers, etc.)
* Patients with central nervous system disease (dementia, stroke, epilepsy, brain tumor, psychiatric disease, etc.)
* Patients who cannot understand the consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2024-04-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between changes in ANI and EEG band power in response to surgical stimulation. | When the laparoscope is inserted
  Correlation between changes in ANI and EEG band power in response to surgical stimulation

SECONDARY OUTCOMES:
Correlation between changes in ANI and EEG band power in response to tracheal intubation | When the tracheal intubation is conducted
  Correlation between changes in ANI and EEG band power in response to tracheal intubation
Correlation between changes in ANI and EEG connectivity in response to surgical stimulation | When the laparoscope is inserted
  Correlation between changes in ANI and EEG connectivity in response to surgical stimulation
Correlation between changes in ANI and EEG connectivity in response to tracheal intubation | When the tracheal intubation is conducted
  Correlation between changes in ANI and EEG connectivity in response to tracheal intubation
Correlation between changes in ANI, EEG band power and NRS in response to analgesic administration | When analgesic drug is administered in the PACU.
  Correlation between changes in ANI, EEG band power and NRS in response to analgesic administration
Correlation between changes in ANI, EEG connectivity and NRS in response to analgesic administration | When analgesic drug is administered in the PACU.
  Correlation between changes in ANI, EEG connectivity and NRS in response to analgesic administration
Differences in EEG band power(Delta, Theta, Alpha, Beta, Gamma) during surgery between groups with large and small changes in ANI | From the beginning of surgery to the end of surgery
  Differences in EEG band power(Delta, Theta, Alpha, Beta, Gamma) during surgery between groups with large and small changes in ANI
Differences in EEG connectivity during surgery between groups with large and small changes in ANI | From the beginning of surgery to the end of surgery
  Differences in EEG connectivity during surgery between groups with large and small changes in ANI
Differences in EEG band power(Delta, Theta, Alpha, Beta, Gamma) during recovery between groups with large and small changes in ANI | From admission to the PACU to discharge from the PACU
  Differences in EEG band power(Delta, Theta, Alpha, Beta, Gamma) during recovery between groups with large and small changes in ANI
Differences in EEG connectivity during recovery between groups with large and small changes in ANI | From admission to the PACU to discharge from the PACU
  Differences in EEG connectivity during recovery between groups with large and small changes in ANI
Differences in EEG band power(Delta, Theta, Alpha, Beta, Gamma) depending on the type of inhaled anesthetic | From the beginning of surgery to the end of surgery
  Differences in EEG band power(Delta, Theta, Alpha, Beta, Gamma) depending on the type of inhaled anesthetic
Differences in EEG connectivity depending on the type of inhaled anesthetic | From the beginning of surgery to the end of surgery
  Differences in EEG connectivity depending on the type of inhaled anesthetic
Differences in ANI depending on the type of inhaled anesthetic | From the beginning of surgery to the end of surgery
  Differences in ANI depending on the type of inhaled anesthetic

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided